CLINICAL TRIAL: NCT01473667
Title: Superficial Cervical Plexus Block for Pacemaker Insertion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in practice occured
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher B. Robards, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11-005969
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Pacemaker Insertion; Regional Block; Pain
MeSH Terms: conditions — Pain | interventions — Urocortins; Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Superficial Cervical Plexus Block (Active Comparator)
  Interventions: Procedure: Superficial Cervical Plexus Block (SCP) block
- Local Infiltration (Active Comparator)
  Interventions: Procedure: Local site infiltration

INTERVENTIONS:
Procedure: Superficial Cervical Plexus Block (SCP) block — SCP block using 10-15ml of 1% Ropivacaine
  Arms: Superficial Cervical Plexus Block
Procedure: Local site infiltration — Local site infiltration using 2% lidocaine
  Arms: Local Infiltration

SUMMARY:
The purpose of this study is to investigate clinical outcomes from two current standard of care pain control procedures performed for patients undergoing pacemaker insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100 years old
* Registered patients at Mayo Clinic in Florida scheduled to undergo primary insertion of pacemaker

Exclusion Criteria:

* Emergency placement of pacemaker
* Sub-pectoral placement of pacemaker
* Patients with history of chronic pain
* Patients with anatomical abnormality or disruption to the pacemaker insertion site or site of block placement
* Patients with allergy to local anesthetic

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To decrease opioid requirements after Pacemaker insertion | first 24 hrs post pacemaker insertion

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Robards, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States